CLINICAL TRIAL: NCT04901442
Title: A Randomised Control Trial to Compare Comfort, Rate of Injury and Speed While Running Using Prefabricated Orthotic Inserted Into Running Shoes vs Running With no Additional Orthotic Inside the Running Shoe
Brief Title: Orthotics and Running
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Talita Cumi Ltd. (Industry)
Collaborators: Aetrex Worldwide Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FFPETFETS001
Record Dates: First submitted 2021-05-14; First posted 2021-05-25 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Running Comfort; Running Speed; Occurence of Running Related Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Running with an Orthotic (Active Comparator): Group A will receive an L700 Speed Orthotic (https://www.aetrex.com/running-orthotic/?lang=en_US) according to participants shoe size and will run with this Orthotic in the participants normal running shoes. The investigators will send an instruction sheet along with the Orthotic in the post, explaining how to use it. Alternatively, an online video tutorial on how to use the Orthotic will also be available throughout the study. The group will be asked to run as normal over the 8-week trial period
  Interventions: Device: Aetrex L700 Speed orthotic
- Running without an Orthotic (No Intervention): Group B will not be provided with the Orthotic and will run in the participants normal running shoes during the course of the study. The group will be asked to run as normal over the 8-week trial period. At the end of the study and following collection of data participants in Group B will also be provided with an L700 Speed Orthotic.

INTERVENTIONS:
Device: Aetrex L700 Speed orthotic — An orthotic insole to be inserted into running shoes. Features Aetrex Arch Support to help biomechanically align the body & help prevent common foot pain such as Plantar Fasciitis, Arch Pain, and Metatarsalgia. Helps prevent injury, alleviate discomfort and helps reduce fatigue while running
  Arms: Running with an Orthotic

SUMMARY:
To investigate whether a prefabricated Orthotic inserted into running shoes will increase comfort, decrease injury and improve speed during recreational running as compared to running shoes without the prefabricated Orthotic.

DETAILED DESCRIPTION:
Running is the most accessible sport in the world. Data from the UK House of Commons has indicated that running has become the favourite exercise among adults 16 or older. However, as the sport grows, so too does the number of running-related injuries (RRIs).

An Orthotic is a device that is placed inside the shoe and functions as a cushion to absorb the shock transmitted on contact with the ground; in addition, they also affect muscle activation that can benefit the user. However, in contemporaneous medical literature, there are mixed views and opinions on whether the use of Orthotics reduces running-related injuries.

This is a randomised control trial that will be conducted over an 8-week period, during which participants will be asked to complete runs and provide data in the form of completed surveys. The primary objective of this study is to investigate whether a prefabricated Orthotic inserted into running shoes will increase comfort, decrease injury and improve speed during recreational running as compared to running shoes without the prefabricated Orthotic.

The study population will include 106 participants who will be randomised into the study and control group. Participants in the study group will be provided with an Orthotic and will run with this in the participants normal running shoes. Participants in the control group will not be provided with the Orthotic and will run in the participants regular running shoes.

All participants (in both groups) will be asked to provide data following each run and also once a week regarding any injury sustained in the preceding 7 days. The minimum required data set will comprise of the personal details and consent on initial enrolment, ongoing consent and data from at least 10 runs (there are 5 individual pieces of information from each run - the date of the run, the distance, the time taken, whether an Orthotic was used or not and the comfort during the run), and injury data every week during the 8 week study period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over.
* Used to running at least 5kms in the last 1 year.

Exclusion Criteria:

* Are currently using a prescription orthotic.
* Have any ongoing pain or deformity in the foot.
* Have been advised by a doctor to not exercise due to a serious health condition.
* Have undergone any surgery in the last 6 months.
* Have undergone any surgery on the foot during lifetime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in levels of comfort as assessed by a Visual Analogue Scale (VAS) | Up to 8 weeks
  Participants will record Comfort on a self-report Visual analogue scale (VAS) of 0 to 10 scale where 0 is "No comfort" and 10 is "Maximum comfort"
Running Duration via a self report questionnaire | Up to 8 weeks
  Participants will record run duration in Hours:Minutes
Running Distance via a self report questionnaire | Up to 8 weeks
  Participants will record run distance in Kilometres/Miles.

SECONDARY OUTCOMES:
Running related Injuries | Once a week during the 8-week trial period.
  Participants will report any running related injuries via a self-report questionnaire. A human model will be used to identify the area of pain. Further choices and information will be provided to the participant on common injuries to allow the identification of the injury. This is a binary measure to observe whether an injury was sustained or not.

CONTACTS AND LOCATIONS:
Overall Officials: George Ampat, MBBS, MS, FRCS, Principal Investigator — Talita Cumi Ltd.
Locations (1):
- Talita Cumi LTD., Southport, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, data will be fully anonymised. Only non-identifiable, anonymised data will be archived along with the publication for use of other researchers. For instance, the age, sex, and study results of participants will be archived indefinitely as a supplementary document to the publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available at the completion of the study on 31/12/2022. It will be available for other researchers indefinitely.
Access Criteria: The non-identifiable data will be openly available as a supplementary document to the publication.

REFERENCES:
- [Background] Collier R. Orthotics work in mysterious ways. CMAJ. 2011 Mar 8;183(4):416-7. doi: 10.1503/cmaj.109-3802. Epub 2011 Feb 14. No abstract available. PMID 21324862
- [Background] Yamato TP, Saragiotto BT, Lopes AD. A consensus definition of running-related injury in recreational runners: a modified Delphi approach. J Orthop Sports Phys Ther. 2015 May;45(5):375-80. doi: 10.2519/jospt.2015.5741. Epub 2015 Mar 26. PMID 25808527
- [Background] Lindorfer J, Kroll J, Schwameder H. Comfort assessment of running footwear: Does assessment type affect inter-session reliability? Eur J Sport Sci. 2019 Mar;19(2):177-185. doi: 10.1080/17461391.2018.1502358. Epub 2018 Jul 25. PMID 30044208
- [Result] van Gent RN, Siem D, van Middelkoop M, van Os AG, Bierma-Zeinstra SM, Koes BW. Incidence and determinants of lower extremity running injuries in long distance runners: a systematic review. Br J Sports Med. 2007 Aug;41(8):469-80; discussion 480. doi: 10.1136/bjsm.2006.033548. Epub 2007 May 1. PMID 17473005
- [Result] Kemler E, Blokland D, Backx F, Huisstede B. Differences in injury risk and characteristics of injuries between novice and experienced runners over a 4-year period. Phys Sportsmed. 2018 Nov;46(4):485-491. doi: 10.1080/00913847.2018.1507410. Epub 2018 Aug 21. PMID 30071170
- [Result] Mundermann A, Stefanyshyn DJ, Nigg BM. Relationship between footwear comfort of shoe inserts and anthropometric and sensory factors. Med Sci Sports Exerc. 2001 Nov;33(11):1939-45. doi: 10.1097/00005768-200111000-00021. PMID 11689747
- [Result] Bonanno DR, Murley GS, Munteanu SE, Landorf KB, Menz HB. Effectiveness of foot orthoses for the prevention of lower limb overuse injuries in naval recruits: a randomised controlled trial. Br J Sports Med. 2018 Mar;52(5):298-302. doi: 10.1136/bjsports-2017-098273. Epub 2017 Oct 22. PMID 29056595
- [Result] Franklyn-Miller A, Wilson C, Bilzon J, McCrory P. Foot orthoses in the prevention of injury in initial military training: a randomized controlled trial. Am J Sports Med. 2011 Jan;39(1):30-7. doi: 10.1177/0363546510382852. Epub 2010 Nov 1. PMID 21041512
- [Result] van der Worp MP, ten Haaf DS, van Cingel R, de Wijer A, Nijhuis-van der Sanden MW, Staal JB. Injuries in runners; a systematic review on risk factors and sex differences. PLoS One. 2015 Feb 23;10(2):e0114937. doi: 10.1371/journal.pone.0114937. eCollection 2015. PMID 25706955
- [Result] Yeung SS, Yeung EW, Gillespie LD. Interventions for preventing lower limb soft-tissue running injuries. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001256. doi: 10.1002/14651858.CD001256.pub2. PMID 21735382
- [Result] Bonanno DR, Landorf KB, Munteanu SE, Murley GS, Menz HB. Effectiveness of foot orthoses and shock-absorbing insoles for the prevention of injury: a systematic review and meta-analysis. Br J Sports Med. 2017 Jan;51(2):86-96. doi: 10.1136/bjsports-2016-096671. Epub 2016 Dec 5. PMID 27919918
- [Result] Ampat, G., R. Baxter, and F. Geoghegan. Pedobarograph based prefabricated orthotics reduces self-reported minor injuries and improves comfort whilst running. MOJ Orthop Rheumatol 12.1 (2020): 1-5.
- See also: Link to government statistics on sports participation in England — https://researchbriefings.parliament.uk/ResearchBriefing/Summary/CBP-8181
- See also: Link to Aetrex website, who produce and provide the orthotic insoles — http://www.aetrex.com/